CLINICAL TRIAL: NCT02755454
Title: Perfusion CT Imaging in Patients With Lung Malignancies Receiving Stereotactic Body Radiation Therapy (SBRT)
Brief Title: Perfusion CT Imaging in Lung Cancer With SBRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-5386-CE
Record Dates: First submitted 2016-03-07; First posted 2016-04-29 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Other): Perfusion CT Imaging
  Interventions: Device: Perfusion CT Imaging

INTERVENTIONS:
Device: Perfusion CT Imaging

SUMMARY:
The goal of this study is to determine specific perfusion patterns for radiation induced lung changes and residual/recurrent lung malignancies in patients treated with stereotactic body radiotherapy SBRT and thus improve to distinguish radiation changes from residual/recurrent lung cancers. Currently CT is often unable to make a clear differentiation between benign and malignant changes in the lung after SBRT treatment necessitating additional wait time to perform follow up CTs or biopsies. Optimal treatment may be delayed. The investigators want to apply a CT perfusion sequence in addition to the routine follow up CTs with the goal to obtain perfusion values of post treatment lung changes and lung tumours. The investigators' hypothesis is that CT perfusion values will help differentiate benign post radiation changes from residual/recurrent tumour in the lung with higher confidence and may help avoid unnecessary delays in cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* CT ordered for baseline and follow up in patients with lung cancer and lung metastases treated with
* Patient will sign a consent form prior to study entry
* Lung cancer and lung metastases are biopsy proven

Exclusion Criteria:

* Patients who are unable to give valid informed consent
* Patients who are unwilling or unable to undergo a CT exam, including subjects with contra-indications to CT exams or intravenous contrast material administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Imaging of during and after SBRT treatment for lung malignancies with a combined perfusion and routine CT to assess therapy response of lung cancer and metastases. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Rogalla, MD, Principal Investigator — UHN
Locations (1):
- Patrik Rogalla, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No